CLINICAL TRIAL: NCT03010852
Title: Focused Incentive Spirometry Monitoring to Reduce Postoperative Oxygen Therapy and Respiratory Complications After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-1268
Record Dates: First submitted 2016-12-07; First posted 2017-01-05 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Respiratory Complication
Keywords: Bariatric Surgery; Spirometry Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care incentive spirometer (No Intervention): Patients in the SOC cohort will not receive the preoperative education and only one postoperative visit per day to collect their self-reported use of IS, if prescribed, and respiratory symptoms but avoiding increasing their awareness of POH, O2 therapy and IS.
- Focused incentive spirometer education and monitoring (Experimental): One of the study investigators will meet eligible patients in the preoperative visit to the UCH Weight Loss Surgery clinic, inform and consent the patient and introduce the first education on IS therapy, highlighting its possible benefits and the importance of compliance (patient's inspiratory effort and frequency). This IS education will be repeated in the preoperative area immediately before surgery. The site will then follow the patient postoperatively. The site will directly check on the patient in the PACU and later in his/her hospital room at least 3 times a day during the first 3 days or sooner if their O2 therapy is discontinued for 2h. During these PO check ups The site will reinforce the IS use, monitor the patient's performance of IS and ask him/her about other respiratory symptoms.
  Interventions: Behavioral: Focused incentive spirometer education and monitoring

INTERVENTIONS:
Behavioral: Focused incentive spirometer education and monitoring
  Arms: Focused incentive spirometer education and monitoring

SUMMARY:
Postoperative (PO) hypoventilation, atelectasis and hypoxemia after bariatric surgery are common and multifactorial, contributing to prolonged oxygen (O2) therapy after surgery and even at hospital discharge. Incentive spirometry (IS) is recommended postoperatively but its success in preventing postoperative atelectasis and hypoxemia (POH) heavily depends on patient compliance with IS effort and frequency. The investigators hypothesize that a focused education preoperatively on IS for POH and intensive monitoring of patient compliance with IS therapy in the early postoperative period shortens postoperative oxygen therapy, decreases POH episodes, and improves respiratory outcomes after bariatric surgery, compared to patients receiving standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients having planned elective bariatric surgery at University of Colorado Hospital

Exclusion Criteria:

* Emergency procedure
* Oxygen therapy within the previous 30 days
* Smoking within the previous 30 days
* Inability or refusal to provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Frequency of at least one episode of moderate/severe hypoxemic event | During first post operative day

SECONDARY OUTCOMES:
Duration of postoperative oxygen therapy | Up to 7 days after surgery
  The duration of postoperative oxygen therapy will be evaluated from the arrival to the post-anesthesia care unit to successful discontinuation of oxygen therapy lasting greater than 2 hours.
Presence of postoperative oxygen therapy and postoperative hypoxemic events | Up to 7 days after surgery
  The development of postoperative hypoxemic events will be evaluated from the initiation of post-operative oxygen therapy through hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Fernandez-Bustamante, M.D., Ph.D., Principal Investigator — University of Colorado, School of Medicine - Department of Anesthesology
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
N/A IPD will not be shared with other researchers